CLINICAL TRIAL: NCT02717858
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Parallel Group Trial to Assess the Effects of Liraglutide on Gallbladder Emptying in Overweight and Obese Subjects
Brief Title: A Trial to Assess the Effects of Liraglutide on Gallbladder Emptying in Overweight and Obese Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-4192; 2014-004772-38 (EudraCT Number); U1111-1163-4641 (Other: WHO)
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Injected s.c./subcutaneously (under the skin) Dose escalation period starting with liraglutide 0.6 mg per day and escalated with weekly increments of 0.6 mg until the target dose 3.0 mg is reached.
  Arms: Liraglutide
Drug: placebo — Injected s.c./subcutaneously (under the skin) once daily.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the effects of liraglutide on gallbladder emptying in overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) equal to or above 27.0 kg/m^2
* Stable body weight (less than 3 kg self-reported change during the previous 3 months)
* Ultrasound assessment of gallbladder volume of an acceptable quality at screening, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or longacting injections))
* History of gastrointestinal surgery or other medical procedure precluding gallbladder emptying assessment (appendectomy is allowed) or any significant digestive disease per the judgement of the investigator
* History of pancreatitis (acute or chronic) or any gallbladder disease (incl. gallstones, gallbladder sludge, or polyps)
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Maximum postprandial gallbladder ejection fraction (GBEFmax) | At 12 weeks (visit 9)

SECONDARY OUTCOMES:
GBEFmax (maximum gallbladder ejection fraction) after first treatment dose | At first treatment dose (visit 4, day 2)
Gallbladder volume | At first dose (visit 4, day2),after 12 weeks (visit 9, day 85)
Gallbladder volume | At 12 weeks (visit 9)
Area under gallbladder EF-time (ejection fraction) curve | At first dose (visit 4, day 2),after 12 weeks (visit 9, day 85)
Area under gallbladder EF-time curve | At 12 weeks (visit 9)
Area under the paracetamol concentration-time curve | At first dose (visit 4,day 2) after 12 weeks (visit 9, day 85)
Area under the paracetamol concentration-time curve | At 12 weeks (visit 9)
Incremental area under the plasma glucose concentration-time curve | At first dose (visit 4,day 2) after 12 weeks (visit 9, day 85)
Incremental area under the plasma glucose concentration-time curve | At 12 weeks (visit 9)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hellerup, Denmark

REFERENCES:
- [Result] Nexoe-Larsen CC, Sorensen PH, Hausner H, Agersnap M, Baekdal M, Bronden A, Gustafsson LN, Sonne DP, Vedtofte L, Vilsboll T, Knop FK. Effects of liraglutide on gallbladder emptying: A randomized, placebo-controlled trial in adults with overweight or obesity. Diabetes Obes Metab. 2018 Nov;20(11):2557-2564. doi: 10.1111/dom.13420. Epub 2018 Jul 10. PMID 29892986
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com